CLINICAL TRIAL: NCT06214325
Title: Music Therapy to Address Patients' Journeys With Chronic Illness, Outcomes, and Readmission
Acronym: MAJOR CHORD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Kulas Foundation (Other)
Responsible Party: Principal Investigator, Samuel Rodgers-Melnick, Integrative Health Research & Data Specialist, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY20230897
Record Dates: First submitted 2024-01-09; First posted 2024-01-19 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Chronic Obstructive Pulmonary Disease
Keywords: Music Therapy; Chronic Obstructive Pulmonary Disease; Heart Failure; In-person; Virtual
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Music Therapy (Experimental): Participants will receive 2 in-person music therapy sessions during hospital admission and 2 virtual music therapy sessions post-discharge.
  Interventions: Behavioral: Music Therapy

INTERVENTIONS:
Behavioral: Music Therapy — Board-certified music therapists (i.e., MT-BC credential) will provide two music therapy sessions, a minimum of 24 hours apart, that include education and disease-specific content (e.g., harmonica exercises for respiratory health [COPD] or music-based breathing exercises [HF]) prior to patients' discharge and two virtual music therapy sessions that address music-assisted relaxation and imagery, additional techniques for managing psychosocial stressors, and gratitude exercises post-discharge.

SUMMARY:
Conduct a pilot study (n = 20) to explore the feasibility and acceptability of the MAJOR CHORD music therapy (MT) intervention (i.e., two in-person MT sessions prior to discharge and two virtual MT sessions post-discharge) and collection of patient-reported outcomes through 30 days after hospital discharge. The investigators will uncover any potential modifications that need to be made to the intervention and data collection process prior to initiating the randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Age range: ≥40 to ≤89 years
* Hospitalized at UH Cleveland Medical Center (UHCMC) with anticipated length of stay following recruitment ≥ 2 days as documented in electronic health record (EHR)
* Diagnosed (i.e., ICD-10 code within the EHR) with either COPD (J44) or HF (I50) with confirmed ICD-10 code in EHR
* Able to read and understand English
* Screening positive for depression and/or anxiety as evidenced by: GAD-7 anxiety score ≥ 10 and PHQ-9 depression score ≥ 10
* Access to WiFi, active email address & laptop, tablet, and/or PC with videoconferencing capabilities
* Has reliable support person who can be available to respond in case of a medical emergency at any time
* Has reliable access to a mobile device with active data plan

Exclusion Criteria:

* Significant hearing and/or visual impairment as documented in EHR
* Unable to independently provide consent (i.e., no proxy consent)
* Active suicidal ideation documented in inpatient psychiatry note during current hospital admission or expressed at any point verbally or in writing to study staff
* Severe psychological comorbidity (e.g., psychosis, schizophrenia) that would prevent patient from engaging fully in intervention as documented in EHR
* Currently admitted to intensive care unit
* Receiving active cancer treatment (e.g., chemotherapy, radiation, immunotherapy) as documented in EHR
* Diagnosed with medical condition likely to be terminal within 24 weeks as documented in EHR
* On wait list for heart transplantation or ventricular assist device (VAD) as documented in EHR
* NYHA Stage IV HF or end-stage COPD as documented in EHR
* Receiving hospice care as documented in EHR
* Active substance abuse as documented in EHR

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
Comparison of actual and anticipated recruitment rates | 30 days post discharge
  Actual rates of recruitment as compared to the anticipated recruitment rate of at least 35% of those approached for the study.
Comparison of actual and anticipated retention rates | 30 days post discharge
  Actual rates of retention as compared to the anticipated retention rate of 70% of participants until the final survey time point.
Comparison of actual and anticipated attendance rates | 30 days post discharge
  Actual rates of attendance rates as compared to the anticipated 3/4 sessions among at least 70% of participants in the music therapy arm.
Comparison of actual and anticipated completion rates | 30 days post discharge
  Actual rates of completion rates as compared to the anticipated at least 70% of 15-day and 30-day follow-up measures.
Number of participants report daily music exercise use | 30 days post discharge
  At least 60% of participants in the music therapy arm reporting use of music exercises at least once every other day.
Acceptance of music therapy intervention | 37 days post discharge
  Favorable responses to qualitative interviews

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Rodgers-Melnick, MPH, MT-BC, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu H, Foss A, Segall TL, Block S, Risser K, Razzak R, Zacharias M, Teba CV, Rodgers-Melnick SN. Refining a hybrid music therapy intervention for chronic obstructive pulmonary disease and heart failure: a single arm pilot study. BMC Complement Med Ther. 2025 Apr 14;25(1):139. doi: 10.1186/s12906-025-04887-x. PMID 40229734